CLINICAL TRIAL: NCT02337842
Title: Phase I Study to Determine the Optimal Human Challenge Dose for a Norovirus GII.4 Challenge Stock (CIN-1)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 12-0033; HHSN272200800006C
Record Dates: First submitted 2015-01-08; First posted 2015-01-14 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2015-08

CONDITIONS: Gastroenteritis Norovirus
Keywords: NoV, CIN-1, GII4. Norovirus, challenge, FUT-2 gene, HBGA-blocking Ab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Cohort 1 (Experimental): N= 9 subjects will receive single oral dose of GII.4 CIN-1 at 10^3 RT-PCR units and N=1 single oral dose Placebo.
  Interventions: Biological: Norovirus GII.4 Challenge Pool CIN-1; Other: Placebo
- Cohort 2 (Experimental): N=9 subjects will receive single oral dose of GII.4 CIN-1 either at 10^2 or 5x10^3 RT-PCR units and N=1 single oral dose of Placebo.
  Interventions: Biological: Norovirus GII.4 Challenge Pool CIN-1; Other: Placebo
- Cohort 4 (Experimental): N=36 subjects will receive single oral dose of GII.4 CIN-1 at either 5x10^4 or 5x10^3 or 10^3 or 10^2 or 10^4 or 5x10^2 or 5x10^1RT-PCR units , N=4 subjects receive a single oral dose of Placebo
  Interventions: Biological: Norovirus GII.4 Challenge Pool CIN-1; Other: Placebo
- Cohort 3 (Experimental): N=18 subjects will receive single oral dose of GII.4 CIN-1 at either 10^4, 10^3, 5x10^2 or 5x10^1 RT-PCR units and N=2 single oral dose of Placebo
  Interventions: Biological: Norovirus GII.4 Challenge Pool CIN-1; Other: Placebo

INTERVENTIONS:
Biological: Norovirus GII.4 Challenge Pool CIN-1 — Norovirus Challenge GII.4 Strain 031693. Cohort 1: receive single oral dose of GII.4 CIN-1 at 10^3 RT-PCR units. Cohort 2: single oral dose of GII.4 CIN-1 either at 10^2 or 5x10^3 RT-PCR units. Cohort 3: single oral dose of GII.4 CIN-1 at either 10^4, 10^3, 5x10^2 or 5x10^1 RT-PCR units. Cohort 4: single oral dose of GII.4 CIN-1 at either 5x10^4 or 5x10^3 or 10^3 or 10^2 or 10^4 or 5x10^2 or 5x10^1RT-PCR units.
Other: Placebo — Placebo: 80 ml of sterile water for oral administration

SUMMARY:
This is phase I, double blind, placebo-controlled safety and infectivity study of experimental human Norovirus genogroup GII.4 administered to healthy adults 18-49 years of age. Subjects susceptible to the human norovirus GII.4 challenge strain. The challenge study will be conducted in 2-3 cohorts of approximately 20 subjects each.Subjects will remain in the inpatient facility for at least four days following challenge and assessed daily for clinical and virologic evidence of norovirus infection. The primary objectives are to evaluate the safety and reactogenicity of the norovirus GII.4 (CIN-1; 031693) challenge stock and to determine a safe and optimal challenge dose of Norovirus GII.4 Challenge Stock norovirus to achieve illness in > /=50% of subjects. Illness is defined as: diarrhea (>3 loose or liquid stools or >300 gm of loose or liquid stool /24h), and/or vomiting during the inpatient period, in a participant with evidence of infection.

DETAILED DESCRIPTION:
This is phase I, double blind, placebo-controlled safety and infectivity study of experimental human Norovirus genogroup GII.4 administered to healthy adults 18-49 years of age. The unblinded pharmacist will assign treatments. Subjects will be admitted to an inpatient nursing unit, challenged with live GII.4 Norovirus strain by oral administration, remain in the unit for at least 4 days following challenge and then followed for post-challenge safety and efficacy with multiple clinical assessments and collection of blood and stool specimens.

Subjects susceptible to the human norovirus GII.4 challenge strain, CIN-1 (i.e. presence of a functional FUT-2 gene), regardless of ABO blood type, will be housed in the Cincinnati Center for Clinical Research (CCCR) inpatient facility and challenged orally with different doses of the virus. The challenge study will be conducted in 2-3 cohorts of approximately 20 subjects each, with the initial cohort receiving 103 RT-PCR units or placebo (9 "challenge" and 1 "placebo" per 10 subjects). Based on the illness rate of acute gastroenteritis (AGE) in the initial cohort, the second cohort will be enrolled to receive a challenge dose based on the results of the previous studies. Additional cohorts may be necessary. Illness is defined as infection accompanied by vomiting and/or diarrhea during the inpatient stay.Two to three additional subjects per cohort will serve as alternates in the event that any of the study subjects are unavailable or become ineligible at the time of the inpatient study.Subjects will remain in the inpatient facility for at least four days following challenge and assessed daily for clinical and virologic evidence of norovirus infection. Subjects will return to the investigational site for evaluation on Day 6 (6-8 days) and about 15 (14-16 days) and 30 days (28-35 days), and 45 (40-45 days), and (55-65) post challenge.

The primary objectives are to evaluate the safety and reactogenicity of the norovirus GII.4 (CIN-1; 031693) challenge stock and to determine a safe and optimal challenge dose of Norovirus GII.4 Challenge Stock norovirus to achieve illness in > /=50% of subjects. Illness is defined as: diarrhea (>3 loose or liquid stools or >300 gm of loose or liquid stool /24h), and/or vomiting during the inpatient period, in a participant with evidence of infection. The secondary objectives are to determine the rate of infection in study participants by; virus detection in stool by Norovirus GII.4 Challenge Stock-specific qRT-PCR and anti- Norovirus GII.4 Challenge Stock serum IgG by ELISA (> /=4 fold rise from baseline to Day 30), determine the quantity and duration of virus shedding in stool by qRT-PCR, conduct Time-to-event analysis to estimate the median time to cessation of shedding using Kaplan-Meier methods, determine the modified Vesikari score as a measure of gastroenteritis severity, determine Norovirus GII.4 Challenge Stock-specific immunoglobulin titers by ELISA before and after the challenge; Serum IgA and IgG, Serum Blockade IgG, Salivary IgA, determine the effect of preexisting Norovirus GII.4 Challenge Stock-specific Immunoglobulin in serum and saliva on the rate of infection, determine total and Norovirus GII.4 Challenge Stock-specific IgA- and IgG-Secreting Cells in circulation by ELISpot assay.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria:

* Subject able to provide written informed consent.
* Male or non-pregnant females between the ages of 18 and 49 years, inclusive.
* Women of childbearing potential must be practicing abstinence or using an acceptable method of birth control for at least 30 days prior to enrollment through day 45 after receipt of the challenge virus. Male subjects must agree not to father a child prior to day 45 after receipt of the challenge virus.

  * A woman is considered of childbearing potential unless post-menopausal (absence of menses for >/= 1 year) or surgically sterilized (tubal ligation, bilateral oophorectomy or hysterectomy).
  * Acceptable contraception methods for women include but are not limited to: sexual abstinence from intercourse with men, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject enrolling in the study, barrier methods such as condoms or diaphragms with spermicide or foam, effective devices (IUDs, NuvaRing®) or licensed hormonal products such as implants, injectables or oral contraceptives.
* For women of childbearing potential, must have a negative serum or urine pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to challenge.
* Are in good general health, as determined by the study investigator within 60 days of challenge.
* Demonstrate knowledge and comprehension of the study by scoring >/=70 procent on a quiz of the study protocol and policies.
* Willing and able to participate in all study visits, including an inpatient stay of at least 96 hours.
* Demonstrated to be secretor positive for HBGA binding.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will be excluded from study participation:

* Have household contact with or have daily contact with children less than 2 years of age or persons older than 70 years of age.
* Have expected occupational or social contact with immunocompromised individuals in the 8 weeks after challenge, including persons with HIV infection or active cancer, children < 2 years of age, pregnant women or persons who are immunosuppressed (e.g. history of stem cell or organ transplantation) and/or provide any child day care services (in-home or non-residential facility).
* Are healthcare workers with patient contact in the 8 weeks after challenge.
* Are food service workers expected to prepare/handle food in the 8 weeks after challenge.
* Plan to be living in a confined environment (e.g. ship, camp, or dormitory) within 8 weeks after receiving the challenge strain.
* For females, are pregnant or plan to become pregnant at any time between the Screening Visit through 45 days after receipt of the challenge virus.
* Are breastfeeding or plan to breastfeed at any given time throughout the study.
* Have a history of gastroenteritis in the 4 weeks prior to challenge or any history of chronic or recurrent diarrhea or vomiting.
* Have a history of malabsorption or maldigestion disorder (e.g. celiac sprue), major gastrointestinal (GI) surgery, irritable bowel syndrome or any other chronic GI disorders that would interfere with the study, including chronic constipation or increased stool frequency.
* Have moderate or severe illness and/or an oral temperature >/=100.4 degre Fahrenheit and/or diarrhea or vomiting within seven days prior to challenge.
* Have a pulse rate less than 55 bpm or greater than 100 bpm. If heart rate is <55 beats per minute and the investigator determines that this is not clinically significant (e.g., athletes) and heart rate increases > 55 beats per minute on moderate exercise (two flights of stairs), subject will not be excluded.
* Have a systolic blood pressure less than 90 mm Hg or greater than 140 mm Hg on two separate measurements (screening and pre-challenge).
* Have a diastolic blood pressure less than 50 mm Hg or greater than 90 mmHg on two separate measurements (screening and pre-challenge).
* Have long-term use (>/=2 weeks) of high-dose oral (>/= 20 mg per day prednisone or equivalent) or parenteral glucocorticoids, or high-dose inhaled steroids for greater than 7 days in the last 6 months.
* Have an autoimmune, inflammatory, vasculitic or rheumatic disease, including but not limited to systemic lupus erythematosus, polymyalgia rheumatic, rheumatoid arthritis or scleroderma.
* Have HIV, Hepatitis B, Hepatitis C infection or untreated latent syphilis.
* Have a seizure disorder.
* Have an active malignancy or history of malignancy (excluding nonmelanotic skin cancer in remission without treatment for more than 5 years) or current use of immunosuppressive or cytotoxic therapy.
* Have positive fecal culture for E. coli O157:H7, Salmonella, Campylobacter, Yersinia, or Shigella, evidence of norovirus in the stool by RT-qPCR or pathogenic ova and parasites detected on microscopic examination at screening.
* Have abnormal screening laboratory test results per laboratory reported normal values and Section 18 Appendix B for white blood cells (WBCs), hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), bilirubin, potassium, sodium, Hemoglobin A1-c (HgbA1-c) and urine protein.
* Serum creatinine greater than 1.1 x ULN
* Alanine aminotransferase (ALT), greater than 1.1 x ULN.
* Have a chronic condition that the study physician feels would pose a threat to participating subjects, including, but not limited to solid organ or stem cell transplantation, diabetes, clinically significant history of immunosuppressive illness, gall bladder disease, heart disease, lung disease, pancreatic disease, renal disease or neurological disease.
* Have abnormal findings on screening electrocardiogram deemed clinically significant by study physician.
* Have ongoing drug abuse/dependence (including alcohol), or a history of these issues within 5 years of enrollment.
* Have a positive urine test for opiates.
* Have any medical, psychiatric, occupational, or behavioral problems that make it unlikely for the subject to comply with the protocol as determined by the investigator.
* Are unwilling to comply with study procedures including abstaining from smoking for the duration of the inpatient portion of the study.
* Have participated in a previous NoV challenge study or NoV vaccine study.
* Have received experimental products within 30 days before study entry or plan to receive experimental products at any time during the study.
* Plans to enroll in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period, including study interventions such as drugs, biologics or devices.
* Plan to donate blood during the course of the study.
* Have received a live vaccine within 30 days before study entry or plan to receive a live vaccine prior to Day 30 of the study.
* Have received an inactivated vaccine within 14 days before study entry or plan to receive an inactivated vaccine prior to Day 14 of the study.
* Have received parenteral immunoglobulin or blood products within 3 months of the study start, or plan to receive parenteral immunoglobulin or blood products within 3 months after receiving the study agent.
* Use of antibiotics within 7 days prior to entry into the inpatient facility.
* Use of any H2 receptor antagonists (e.g., Tagamet, Zantac, and Pepcid), proton pump inhibitors (e.g., Prilosec, OTC, Protonix, and Prevacid), or prescription acid suppression medication or over-the-counter (OTC) antacids in the 72 hours prior to NoV challenge.
* Use of prescription and OTC medications containing acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs within 48 hours prior to NoV challenge.
* Regular use of laxatives or anti-motility agents.
* Have a history of allergy to sodium bicarbonate.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing any mild, moderate or severe reactogenicity outcomes. | Day 1 to Day 180
Proportion of subjects with Norovirus-GII.4 Challenge Stock (CIN-1; 031693) associated illness following norovirus GII.4 challenge | Day 1 to Day 5
Number of serious adverse events related to virus challenge reported at any point during the study | Day 1 to Day 180
Number of subjects experiencing Grade 3 adverse events after virus challenge throughout the study to day 30 | Day 1 to Day 30
Determine Infectious Dose50 based on infection rate after challenge with various doses. | Day 1 to Day 180

SECONDARY OUTCOMES:
Infection rate within each dose, defined as proportion of subjects excreting challenge virus in stool 24 hours after challenge | 24 hours after challenge
Proportion of subjects with norovirus specific IgG-ASC / 10^6 PBMC (freshly isolated PBMCs) | Day 1 to Day 45
Clinical Severity Score of vomiting and/or diarrhea related to the challenge strain using the Modified Vesikari Scale | Day 1 to Day 5
95% confidence intervals of vomiting and/or diarrhea related to the challenge strain | Day 1 to Day 5
Mean duration (hours) of vomiting and/or diarrhea related to the challenge strain | Day 1 to Day 5
At any time after challenge Proportion of subjects with >/= 4 fold rise from the baseline in virus-specific antibody titers in serum(IgA, IgG Blockade), or salivary IgA | Day 1 to Day 45
Infection rate within each dose defined as proportion of subjects showing a > /=4 fold rise in virus specific serum IgG from baseline to Day 30 | Day 1 to Day 30
Proportion of subjects with norovirus specific IgA- ASC / 10^6 PBMC (freshly isolated PBMCs) | Day 1 to Day 45
Correlation of challenge outcome (infection) and preexisting serum immunoglobulins. | Day 1 to Day 45
Time-to-cessation of virus shedding in stool in hours for each challenge dose. | Day 1 to Day 60
Magnitude and duration of virus shedding in stool reported as qRT-PCR units for each challenge dose | Day 1 to Day 60

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio, United States